CLINICAL TRIAL: NCT03067662
Title: Efficacy of Supervised Physical Exercise in Metabolic Control of Women With Gestational Diabetes
Brief Title: Aerobic Exercise in Women With Gestational Diabetes
Acronym: GDM-FIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Paolo Moghetti, Associate Prof., Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2152
Record Dates: First submitted 2017-02-03; First posted 2017-03-01 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised exercise intervention (Experimental): Women in the intervention group will perform low intensity aerobic exercise three times per week at 30% HRR (Heart Rate Reserve), under continuous heart rate monitoring. Duration of each session will progress from 26 minutes the first week to 40 minutes (by increasing 2 min/week).
  Interventions: Other: Aerobic exercise
- Current standard of care (No Intervention): Women in the control group will receive standard physical exercise recommendations.

INTERVENTIONS:
Other: Aerobic exercise
  Arms: Supervised exercise intervention

SUMMARY:
A few, small randomized controlled trials have investigated the effects of exercise on blood glucose levels in women with gestational diabetes (GDM), with inconsistent results.

To assess the effects of supervised exercise in women with GDM, 48 women with gestational diabetes, diagnosed between the 18th and 28th week of gestation, will be recruited, after exclusion of subjects with contraindications to exercise. These subjects will be randomly assigned to two groups: structured exercise intervention or standard care.

Women in the intervention group will perform low intensity aerobic exercise three times per week at 30% HRR (heart rate reserve), under continuous heart rate monitoring. Duration of each session will progress from 26 minutes the first week to 40 minutes (increasing 2 min/week). Women in the control group will receive standard diet and physical exercise recommendations.

In all women, clinical, metabolic and anthropometric features will be assessed before, during and at the end of the study. Newborn data will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy,
* Gestational diabetes diagnosis between 18th and 28th week of gestation,
* Caucasian.

Exclusion Criteria:

* Hemodynamically significant heart disease,
* Restricted lung disease,
* Incompetent cervix/cerclage,
* Persistent second or third trimester bleeding,
* Placenta previa,
* Threatened preterm labor,
* Ruptured membranes,
* Preeclampsia,
* Hypertension,
* Severe anemia,
* Cardiac arrhythmias,
* History of epilepsy,
* Chronic bronchitis,
* Orthopedic limitations,
* Overt hyperthyroidism/ hypothyroidism,
* Type 1 diabetes mellitus,
* Drugs that interfere with metabolic control (such as cortisone)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-09-27; Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in fasting plasma glucose levels (mg/dL) | Before intervention and at 35-37 week of gestation

SECONDARY OUTCOMES:
Change in body weight (kg) | Before intervention and at 35-37 week of gestation
Change in body mass index (kg/m^2, weight in kilograms, height in meters) | Before intervention and at 35-37 week of gestation
Change in blood pressure (mmHg) | Before intervention and at 35-37 week of gestation
Change in heart rate (HR, beats per minute) | Before intervention and at 35-37 week of gestation
Dosage of insulin therapy, if required | Before intervention and at 35-37 week of gestation
  Insulin units and week at start
Change in caloric intake | Before intervention and at 35-37 week of gestation
  By 3 day-food recall questionnaire (kcal/die)
Change in energy expenditure through voluntary physical activity | Before intervention and at 35-37 week of gestation
  Energy expenditure is estimated by International Physical Activity Questionnaire (IPAQ)
Compliance (percentage) | Throughout the intervention period, an average of 3-5 months according to the gestational week of inclusion in the study
  Attendance at the scheduled sessions is recorded for each patient
Circulating c-reactive protein (CRP) levels (mg/dL) | Before intervention and at 35-37 week of gestation
Adiponectin levels (μg/mL) | Before intervention and at 35-37 week of gestation
Pulse wave velocity (PWV, m/s) | Before intervention and at 35-37 week of gestation
  A non-invasive assessment of arterial stiffness (in the carotid-radial and carotid-femoral parts of the arterial tree) by the technique of applanation tonometry
Quality of life (questionnaire) | Before intervention and at 35-37 week of gestation
  Measured by SF-36 (36-item Short Form Health Survey-36) questionnaire
Depression state (questionnaire) | Before intervention and at 35-37 week of gestation
  Measured by Center of Epidemiological Studies Depression Scale
Glucose concentration during and after exercise | At 32-34 week of gestation
  A continuous glucose monitoring system (CGMS) will be applied at 32-34 week of gestation, and blood glucose will be recorded every 5 min over the following five days. Glucose concentrations during the 40-min exercise session, the subsequent night, and the 24-h period following exercise, as well as during the corresponding periods of a non-exercise day will be recorded, and glucose variability and time spent in hypoglycemia or hyperglycemia will be calculated
Fetus bi-parietal diameter (cm) | At 20, 30, 34-37 week of gestation
Fetus head circumference (cm) | At 20, 30, 34-37 week of gestation
Fetus abdominal circumference (cm) | At 20, 30, 34-37 week of gestation
Fetus femur length (cm) | At 20, 30, 34-37 week of gestation
Weight (kg) of child at birth | 3 months after delivery
Length (cm) of child at birth | 3 months after delivery
Apgar index (score) at 1st and 5th minutes | Birthday
Gender (M/F) | 3 months after delivery
Malformations and neonatal diseases (YES/NO) | 3 months after delivery
Type of delivery (spontaneous, induced, caesarean section) | 3 months after delivery
Week of delivery (wk) | 3 months after delivery
Type of feeding (breastfeeding or bottle feeding) | 3 months after delivery
Weight (kg) of child 3 months after delivery | 3 months after delivery
Length (cm) of child 3 months after delivery | 3 months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Moghetti, MD, PhD, Principal Investigator — University of Verona and Azienda Ospedaliera Universitaria Integrata of Verona
Locations (1):
- Endocrinology, Diabetes and Metabolism Section, Department of Medicine, University of Verona and Azienda Ospedaliera Universitaria Integrata of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No